CLINICAL TRIAL: NCT01991262
Title: A Nationwide Epidemiological, Non-Interventional Study Evaluating an Educational Support Program for Improving Treatment Adherence in Patients With Hepatitis B Viral Infection
Brief Title: A Nationwide Epidemiological, Educational Support Program for Improving Treatment Adherence in Patients With HBV
Acronym: Help-B
Status: Withdrawn | Type: Observational
Why Stopped: the support group need to have some change
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eli Zuckerman, Director of Liver Unit, Carmel Medical Center
Other Study IDs: CMC-13-0112-CTIL
Record Dates: First submitted 2013-11-17; First posted 2013-11-25 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: HBV Treatment Adherence by Support Program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1 phone call and SMS reminder.: cloosed no one enrolled
- Group 2 phone call only.: cloosed no one enrolled
- Group 3 SMS reminder only .: cloosed no one enrolled
- Group 4 (Control) no support: cloosed no one enrolled

SUMMARY:
Protocol Title: A Nationwide Epidemiological, Non-Interventional Study Evaluating an Educational Support Program for Improving Treatment Adherence in Patients with Hepatitis B Viral Infection

Objective(s): The primary objectives of the study are to assess:

* HBV treatment adherence rate in patients enrolled in the Support Program
* Adherence rates at 6m, 12m.

The secondary objectives are to assess:

* Adverse events rate and profile.
* Actual treatment duration and dose taken vs. prescribed.
* The impact of SMS reminders.

Study Design: Eligible patients will be randomized into one of four groups: Group 1 shall receive both a weekly phone call from a supporter and a daily SMS reminder. Group 2 will receive a weekly phone call only. Group 3 will receive a daily SMS reminder only and group 4 (Control) shall receive no support.

Study Population: Adult newly diagnosed with Hep B patients, eligible to begin treatment with first line therapy.

Data Collection Methods:

1. Supporter's documentations of patient's self assessment.
2. Drugs dispense data from pharmacies
3. Pills count.

DETAILED DESCRIPTION:
Protocol Number: AI463-972 Date: 23-Oct-2013 Ver: 2 Observational Study Protocol AI463-972 - Help-B

A Nationwide Epidemiological, Non-Interventional Study Evaluating an Educational Support Program for Improving Treatment Adherence in Patients with Hepatitis B Viral Infection

Prof. Eli Zuckerman; Dr. Yoram Menachem; Prof. Rifat Safadi; Prof. Assy Nimer; Dr. Rawi Hazzan; Dr. Michal Carmiel

Treatment for Chronic HBV The objectives of HBV therapy are to improve upon the spontaneous rates of sustained disease remission (as defined by long-term HBeAg and HBsAg seroconversion rates off-treatment), thereby reducing the risk of disease progression, with resultant improvements in quality of life and reductions in healthcare costs. Seven drugs are presently approved in the USA and/or EU for the treatment of CHB in patients with HBeAg-positive and -negative disease. They fall into 2 classes: antiviral/immunomodulators (IFNα and pegIFNα-2a) and antiviral nucleos(t)ide analogs (NUCs).

EASL and AASLD Treatment Guidelines (2009) recommend that HBV therapy may be initiated with any of the currently approved agents, but that IFNα (standard or pegylated), Tenofovir (TDF) or Entecavir (ETV) are preferred first-line options for treatment of CHB patients with HBeAg-positive and HBeAg-negative disease.

Poor adherence to therapy is a complex challenge for physicians treating patients with chronic diseases. In clini¬cal practice, adherence rates averages 50%, falling most dramatically after the first 6 mo of treatment. Guidelines on CHB therapy emphasise the need for optimal adherence, with risk of resistant viral strains emerging if the virus has a drug free holiday. For example, antiviral resistance has been reported in up to 70% patients after 4 years on Lamivudine, 29% after 5 years of Adefovir dipivoxil and 1% after 4 years of Entecavir monohydrate. The number of dose omissions that may lead to this is variable but any omission poses a po¬tential risk of viral replication breakthrough. Although, the data for CHB are lacking, it is evident from the HIV literature that near-perfect adherence (> 95% adherence rates) is needed to achieve a non detectable viral load and avoid emergence of resistant strains. Hence, in the clinical setting of CHB therapy, the goal of adherence remains 100%.

Unlike other chronic conditions, the rapid viral rep¬lication potential and mutation rates of hepatitis B virus require very high levels of adherence to achieve and maintain virological suppression. Suboptimal adher¬ence risks exacerbating existing liver disease, which can be life-threatening particularly in patients with advanced cirrhosis. Furthermore, it can lead to the development of drug-resistant strains, limiting therapeutic options and additionally poses the public health risks of transmission of drug-resistant viral strains to non-immune individuals in the community, or to those whose previous vaccina¬tion are no longer protective. Given the global burden of the disease, widespread transmission of drug-resistant strains may have serious and wide-reaching consequences.

1.1 Study Rationale Non- adherence to treatment is a well known issue across many therapeutic areas. In Hep C, literature review shows that adherence in real life may reach 65%, with most drop-outs during first 3 months, mainly due to minor side effects. In Hep B, reported adherence studies show 50%-80% adherence, with an average of ~65%. Most drop-outs are during first 6 months of treatment. Non-adherence to treatment is believed to contribute not only to liver deterioration but also to emerging viral resistance.

Studies for adherence support show an average improvement of around 10%-15% at the best. Assessed methods are:

* Patient education
* Patients empowerment
* SMS reminders
* Pills' boxes with electronic reminders

The lack of symptoms along with chronicity of treatment, financial burden and lack of patient's education - are recognized as important factors for non-adherence.

The abundance of new drugs for viral hepatitis, high disease prevalence and the close relation between effective treatment and clinical outcomes - create a clear need for not only providing treatment but also an efficient support system aimed at supporting patients' adherence.

1.2 Research Question We expect that an ongoing patients' support system will contribute to adherence increase. The support should be provided by HCPs, be continuous and provide reminders, medical education and direct contact between patients and HCPs.

Therefore, study hypothesis is:

* An ongoing 6 months adherence support will increase adherence rates for Hep B patients
* Adherence rate increase will be at least 20%.
* Direct weekly telephone contacts will contribute major improvement. Smart phone application daily reminders will contribute as well and there is need to assess its relative contribution.

  2 OBJECTIVES 2.1 Primary Objectives At least 20% improvement in adherence rates for newly treated Hep B patients. Adherence rate will be defined as the per cent of days the patients took their hepatitis B virus medications during study treatment and the number of missed doses.

2.2 Secondary Objectives

The difference in adherence improvement among 3 types of adherence support:

1. Weekly telephone call + daily text messages reminders.
2. Weekly telephone calls.
3. Daily text messages reminders.
4. Control - no adherence support

3 STUDY DESIGN 3.1 Overview of Study Design This is an epidemiological non-interventional study conducted in the community. Medical students (Hereinafter "Supporters"), attending senior years (4th or 5th year) will receive training about the Educational Support Program. In case not all vacancies can be filled with suitable medical students, senior years nursing students will be approached. Every supporter will be supporting a maximum of 10 recruited patients simultaneously. Every 5 supporters will report to a nurse. Every 2 nurses will report to a Hepatologist (Hereinafter "Investigator"). Overall, every Hepatologist shall be recruiting a maximum of 100 patients.

During the pre-study phase, eligible patients, who are prescribed with HBV treatment with Entecavir by their respective Investigator, will be informed of the Support Program. Interested patients will receive ICF for signature. Upon signature, the recruiting Investigator will randomize the newly recruited patient into one of the four study groups.

Randomization will be provided by CHS computerized system (Randomization engine).

Patients in the supported groups (Groups 1; 2 and 3) shall undergo the procedure described hereby:

Upon recruitment, the patient will be introduced to the nurse, who will appoint a supporter to the patient, install the smart-phone reminder application (to relevant groups - Group 1 and Group 3) and explain the support format according to patient's group:

Group 1:

Receive weekly phone calls from their supporters who will monitor HBV treatment adherence and adverse events, respond to the patients' queries, suggest possible remedies to patients' basic complaints (per definition and qualification in training), refer more complex queries and/or complaints to respective nurse and refer patients to physicians for further treatment, if required. The Supporter will record the data on a Patient Follow-Up Form and report, on a monthly basis, to the respective nurse. In addition, patients in this group will install the reminder application on their smart-phones and will be reminded on a daily basis, by the application, to take their medication.

Group 2:

Receive weekly phone calls from their Supporters who will monitor HBV treatment adherence and adverse events, respond to the patients' queries, suggest possible remedies to patients' basic complaints (per definition and qualification in training), refer more complex queries and/or complaints to respective nurse and refer patients to physicians for further treatment, if required. The Supporter will record the data on a Patient Follow-Up Form and report, on a monthly basis, to the respective nurse.

Group 3:

Patients in this group will install the reminder application on their smart-phones and will be reminded on a daily basis, by the application, to take their medication.

Group 4:

Patients in the 4th group (control group) will continue the SOC without any further support.

Every month, patients will receive a letter from their respective Investigators, summarizing their study status in the previous month (Appendix A). Every quarter (3 months), each nurse will report study progress to responsible Investigator and schedule a follow-up appointment for the patient with the investigator. The patient will bring the pill boxes to the follow-up appointment for counting.

At the end of the supporting phase, the patients will continue HBV treatment according to standard care and their physician's instructions. During the follow-up phase, all groups will be handled as Group 4 patients.

3.2 Study Population

Approximately 250 Naïve Hep B patients are expected to participate in the study and will be divided into 4 study arms:

Group 1: 63 pts receiving weekly telephone contact & daily text messages for 6 months.

Group 2: 63 patients receiving weekly telephone contacts for 6 months. Group 3: 63 patients receiving daily text messages for 6 months. Group 4: 63 patients receiving no adherence support.

3.2.1 Inclusion Criteria

* Adult male and female patient (> 18 years).
* Prescribed treatment of Entecavir for HBV
* Must have access to a smart-phone.
* Written informed consent.

3.2.2 Exclusion Criteria

* Patients with hepatitis C, hepatitis D or HIV co-infection.
* Co-infected patients who require additional medication.
* Patients with prior liver transplantation
* Patients with impaired renal function requiring dialysis
* Immune-suppressed patients receiving HBV antiviral prophylaxis
* Pregnant patients.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* Parallel participation in another clinical trial.
* Patients who cannot take medication independently.

3.3 Data Source/Data Collection Process

Adherence to treatment will be assessed by 3 methods:

1. Supporters' weekly documentations.
2. Pill count - Patients will be instructed to bring the boxes to quarterly follow-up visits with the Hepatologist.
3. Drugs dispense data from pharmacies - every 3 months.

Safety assessment will be completed by:

1. Supporters' weekly documentations.
2. Documentation by treating hepatologists, during ongoing visits. 3.4 Definitions of Study Variables Adherence will be quantified into percentage and will be calculated as the percent of days in which the patient took the prescribed medication out of the number of days the patient was instructed to take the medication by prescription.

3.4.1 Outcomes/Endpoint Variables

Primary endpoint:

Adherence rate will be defined as the percentage of days the patients took their hepatitis B virus medications during study treatment and the number of missed doses. Adherence will be measured as a combination of:

1. Drug dispense at pharmacy (every month)
2. Self report by patient (every week)
3. Pills count (every 3 months)

A responder will be defined as a patient with at least 80% adherence to drug treatment.

Secondary endpoint:

The difference in adherence improvement among 3 types of adherence support

1. Weekly Phone Call + Daily Application Reminder
2. Weekly Phone Call
3. Daily Application Reminder

4 STATISTICAL ANALYSIS 4.1 Statistical Analysis Methods All measured variables and derived parameters will be listed individually and, if appropriate, tabulated by descriptive statistics.

For categorical variables summary tables will be provided giving sample size, absolute and relative frequency and 95% CI (Confidence Interval) for proportions by study arm.

For continuous variables summary tables will be provided giving sample size, arithmetic mean, standard deviation, coefficient of variation (if appropriate), median, minimum and maximum, percentiles and 95% CI (Confidence Interval) by study arm for means of variables.

4.1.1 Primary Objective Responders will be defined as patients with at least 80% adherence to drug treatment. 95% Confidence Interval (95% CI) will be calculated for the rate of responders per study arm (arms 1, 2 and 3).

4.1.2 Secondary Objectives Chi-square test or Fisher's Exact test (as is appropriate) will be applied for testing the statistical significance of the difference in responders rate between study arms 1 (Weekly Phone Call + Daily Application Reminder), 2 (Weekly Phone Call) and 3 (Daily Application Reminder) vs. group 4 (no support).

The effect of telephone call will be tested comparing groups 1+2 vs. groups 3+4.

The effect of daily SMS will be tested comparing groups 1+3 vs. group 2+4. Logistic Regression model will be applied for testing the statistical significance of the difference in responders' rate between study arms 1, 2 and 3 vs. group 4 and between the active groups with adjustment to suspected confounders related to study outcome which will be found different between the arms.

Logistic regression will be applied for analyzing the effect of telephone call and daily SMS (as described above) with adjustment to suspected confounders.

All tests will be two-tailed, and a p value of 5% or less will be considered statistically significant.

The data will be analyzed using the SAS ® version 9.1 (SAS Institute, Cary North Carolina).

4.2 Power/Sample Size Rational for Sample size calculation Sample size calculation is based on demonstrating a difference of at least 21% in response rate in the comparison between study arms 1, 2 and 3 vs. group 4. This difference reflects an odds ratio of 0.23 with statistical significance of 5% with statistical power of 80% when the sample size is 252, 63 in each study arm.

Sample Size Justification A two group continuity corrected Chi square test with a 0.050 two-sided significance level will have 80% power to detect the difference between a Group 1 proportion and a Group 2 proportion (odds ratio of 0.231) when the sample size in each group is 64.

Reference: nQuery advisor 2.1

5 STUDY CONDUCT This study will be conducted in accordance with International Society for Pharmacoepidemiology (ISPE) Guidelines for Good Pharmacoepidemiology Practices (GPP) and applicable regulatory requirements.

5.1 Ethics Committee Review and Informed Consent

5.1.1 Ethics Committee Review The investigator must ensure that the required approvals from Ethics Committees, Independent Review Committees, Regulatory Authorities, and/or other local governance bodies are obtained before study initiation at the site.

5.1.2 Informed Consent In accordance with local regulations, subjects should provide either written or oral consent before enrollment into the study. Investigators must ensure that patients, or, in those situations where consent cannot be given by patients, their legally acceptable representatives, are clearly and fully informed about the purpose of the study, potential risks, the patient's rights and responsibilities when participating in this study. If local regulations do not require an informed consent document to be signed by the patient, the site staff should document key elements of the informed consent process in the patient's chart.

This study does not require that informed consent is obtained from patients.

5.2 Responsibilities within the Study The study shall be conducted as described in this approved protocol. All revisions to the protocol must be discussed with, and be prepared by BMS.

5.3 Confidentiality of Study Data The confidentiality of records that could identify patients within the database must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

For the purposes of protecting a patient's identity, a unique code will be assigned to each patient, such as a series of numbers and/or letters (for example, CA180330-0001-00001). The data that is recorded with the patient's assigned code is called "key-coded data". Key-coded study data will be managed by the sponsor and/or its delegates in a study-specific electronic database (the "study database"). Only the investigator and the site staff have access to the link between patient's assigned code and the patient's identity. However, in case of an audit or inspection, subject to local laws and regulations, government officials, IRB/EC representatives and sponsor representatives may access this information at the study site. If the study requires on-site monitoring, subject to local laws and regulations, sponsor representatives will also access the primary data source at the study site (see section 6.4). Data that could directly identify the patient will not be collected in the "study database".

5.4 Quality Control Power/Sample Size Representatives of BMS and/or its delegates must be allowed to visit all study site locations to assess the data quality and study integrity. On site, they will review study files and, if allowed by local laws and regulations, patient medical charts to compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable.

In addition, the study may be evaluated by BMS internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities, and promptly forward copies of inspection reports to BMS.

5.5 Database Retention and Archiving of Study Documents The investigator must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period specified by the sponsor, whichever is longer. The investigator must contact BMS prior to destroying any records associated with the study. Location of database and supporting documentation will be outlined in the final observational study report.

6 ADVERSE EVENT REPORTING The INSTITUTION/PRINCIPAL INVESTIGATOR must notify BMS with the related and non-related Serious Adverse Events (SAEs) and/or Pregnancies within 24 hours of becoming aware of the event.

The INVESTIGATOR must notify BMS with the related and non-related non-serious Adverse Events within 7 days of becoming aware of the event.

All Adverse Events and/or Serious Adverse Events must be reported to:

Bristol-Myers Squibb Company Global Pharmacovigilance FAX Number: 609-818-3804 or Email: WorldWide.Safety@bms.com

The INVESTIGATOR must notify BMS with all Adverse Events in aggregate in the Final Study Report (FSR).

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patient (> 18 years).
* Prescribed treatment of Entecavir for HBV
* Must have access to a smart-phone.
* Written informed consent.

Exclusion Criteria:

* • Patients with hepatitis C, hepatitis D or HIV co-infection.

  * Co-infected patients who require additional medication.
  * Patients with prior liver transplantation
  * Patients with impaired renal function requiring dialysis
  * Immune-suppressed patients receiving HBV antiviral prophylaxis
  * Pregnant patients.
  * Inability or unwillingness to provide informed consent or abide by the requirements of the study.
  * Parallel participation in another clinical trial.
  * Patients who cannot take medication independently.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult newly diagnosed with chronic hepatitis B patients, eligible to begin treatment with first line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hepatitis B treatment adherence rate in patients with support system | 6 months